CLINICAL TRIAL: NCT00548314
Title: Application of a Dermal Substitute and Topical Negative Pressure to Improve the Healing of Burn Wounds
Brief Title: Dermal Substitute and Topical Negative Pressure in Burns
Acronym: VAC-M
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Responsible Party: Association of Dutch Burn Centres, Association of Dutch Burn Centres
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07.109
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Burns
Keywords: Matriderm; Dermal matrix; VAC therapy; Split skin graft; Burns; Scar quality
MeSH Terms: conditions — Burns | interventions — matriderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): After excision and adequate hemostasis, the selected wound will be treated with the dermal substitute Matriderm, a split skin graft (SSG), mesh 1:1.5 and VAC therapy. The VAC system will be set at 125mmHg, continuous mode, for 3-5 days.
  Interventions: Other: dermal matrix; Device: VAC therapy (KCI)
- 2 (Experimental): After excision and adequate hemostasis, the selected wound will be treated with the dermal substitute Matriderm, a split skin graft (SSG), mesh 1:1.5.
  Interventions: Other: dermal matrix
- 3 (Experimental): After excision and adequate hemostasis, the selected wound will be treated with a split skin graft (SSG), mesh 1:1.5 and VAC therapy. The VAC system will be set at 125mmHg, continuous mode, for 3-5 days.
  Interventions: Device: VAC therapy (KCI)
- 4 (Active Comparator): After excision and adequate hemostasis, the selected wound will be treated with a split skin graft (SSG), mesh 1:1.5.
  Interventions: Procedure: Split skin graft

INTERVENTIONS:
Other: dermal matrix — 1mm thickness matrix composed of collagen-elastin hydrolosate
  Other Names: Matriderm
  Arms: 1; 2
Procedure: Split skin graft
  Arms: 4
Device: VAC therapy (KCI) — VAC therapy for 3-5 days 125mmHg
  Arms: 1; 3

SUMMARY:
The purpose of this study is to determine whether a treatment of full thickness wounds by the dermal substitute Matriderm, split skin graft and VAC treatment will improve scar quality, demonstrated by a significant increase of skin elasticity parameters after 3 months.

Additionally, an increase of the take of graft and improvement of scar assessment scale, scar colour/pigmentation and time to complete wound closure, is expected.

DETAILED DESCRIPTION:
The standard therapy for full thickness wounds is transplantation with a split thickness skin graft. However, scars usually develop as a result of this therapy. Previous research has demonstrated an improvement of scar quality if a dermal substitute was applied in combination with a split skin graft in reconstructive wounds, but not so much in burn wounds. One of the problems in burn wounds was the retarded outgrowth of the skin graft when a dermal substitute was applied in a one step procedure with the graft. Since then, application of topical negative pressure has demonstrated that the take and outgrowth of a skin graft can be improved by this technique. It now seems feasible to combine these two technologies in order to improve the quality of healing of burn wounds in the acute phase of healing.

Aim of the study is to investigate if application of a dermal substitute in combination with topical negative pressure can improve the quality of the scar in burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 yrs with acute burns/trauma wounds that require skin grafting
* Minimal study wound surface 10 cm2
* Maximal study wound surface 300 cm2
* Maximal TBSA 15% full thickness wounds
* Informed consent

Exclusion Criteria:

* Patients with wounds without adequate possibility to apply VAC
* Immunocompromised patients
* Infected wounds
* Pregnant patients
* Patients who are expected (according to the responsible medical doctor) to be non-compliant to the study protocol. This includes patients with severe cognitive dysfunction/impairment and severe psychiatric disorders (e.g. borderline or depression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
skin elasticity parameters (representing scar quality) | after 3 months

SECONDARY OUTCOMES:
take of graft after 5-7 days, time to complete (>95%) healing, scar assessment scale and scar colour/ pigmentation (Dermaspectrometer) | after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Esther Middelkoop, Professor, Study Director — Association of Dutch Burn Centres (ADBC)
Locations (1):
- Red Cross Hospital, Beverwijk, North Holland, Netherlands